CLINICAL TRIAL: NCT02657993
Title: Hypnosis to Reduce Aromatase Inhibitor (AI) Associated Musculoskeletal Pain and to Improve AI Adherence: An RCT to Explore Efficacy and Cost Effects
Brief Title: Hypnosis to Reduce Aromatase Inhibitor Pain and Improve Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Guy Montgomery, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 14-1344; R01AT008762-01 (NIH)
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Breast Neoplasms; Musculoskeletal Pain
Keywords: Breast Neoplasms; Aromatase Inhibitors; Musculoskeletal Pain; Hypnosis; Medication Adherence; Cost-Benefit Analysis; Treatment Outcomes
MeSH Terms: conditions — Breast Neoplasms; Musculoskeletal Pain; Medication Adherence | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypnosis (Experimental): The hypnosis intervention involves three, face-to-face, hypnosis sessions delivered by doctoral-level psychology professionals
  Interventions: Behavioral: Hypnosis
- Attention Control (Non-Hypnosis) (Active Comparator): The attention control intervention is matched to the hypnosis intervention in terms of the amount of professional time received by patients.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Hypnosis — The hypnosis intervention involves three parts. First, participants will receive three, face-to-face hypnosis sessions delivered by doctoral-level psychology professionals. The sessions are based on materials developed by experienced psychologists in the Integrative Behavioral Medicine Program at the Icahn School of Medicine at Mount Sinai. Second, participants will be taught how to use hypnosis themselves (self-hypnosis) to help manage their pain. Third, participants will receive a hypnosis recording to listen to in-between sessions and throughout the course of the study. At home hypnosis practice will be recommended.
  Participants will be asked to complete questionnaires over a period of 12 months.
  Arms: Hypnosis
Behavioral: Attention Control — The attention control intervention involves three face-to-face meetings with a doctoral-level psychology professional. During these sessions, participants will be asked to discuss with the interventionist their experience of taking aromatase inhibitors and associated musculoskeletal pain. The interventionist will not lead the patient in imagery, relaxation, evaluation of thought processes, or even simple discussion. Rather interventionists will allow the patient to direct the flow of the conversation and will provide support and empathy. Interventionist contact time in AC sessions will be identical to that in the hypnosis group. Overall, the attention control intervention will control for professional attention.
  Participants will be asked to complete questionnaires over a period of 12 months.
  Other Names: Non-Hypnosis
  Arms: Attention Control (Non-Hypnosis)

SUMMARY:
The purpose of this study is to determine whether hypnosis is efficacious in reducing musculoskeletal pain in breast cancer survivors taking aromatase inhibitors, and by doing so, whether hypnosis can help survivors to be more adherent to their medication regimen.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the efficacy of hypnosis for reducing musculoskeletal pain (MSP) in women taking aromatase inhibitors (AIs) for breast cancer. Research indicates that AIs are associated with musculoskeletal pain in up to 61% of breast cancer survivors. AI-associated MSP can include joint pain in the wrists, hands, and knees; carpal tunnel syndrome and trigger finger; and decreased grip strength, morning stiffness, and general muscle pain. MSP can lead to difficulty performing daily activities and can reduce quality of life in breast cancer survivors. This pain is not only aversive in and of itself, but also is associated with non-adherence to prescribed, daily AI regimens. In some studies, AI non-adherence estimates were as high as 50%.

At the present time, there is no "gold standard" treatment for AI-associated MSP. What is needed is an intervention that: reduces breast cancer survivors' MSP and helps them be more adherent to their prescribed AI regimen, does not have side-effects of its own, does not place a large time or financial burden on survivors, and which can be taught to survivors to practice on their own.

Hypnosis, a mind-body intervention, has been widely demonstrated to reduce pain. In fact, analgesia is perhaps the best known effect of hypnosis. Meta-analyses have consistently supported the efficacy of hypnosis for pain control, including chronic pain. Hypnosis also has a long tradition in cancer symptom management, especially for pain reduction. Hypnosis has been defined as an agreement between a person designated as the hypnotist (e.g., health care professional) and a person designated as the client or patient to participate in a psychotherapeutic technique based on the hypnotist providing suggestions for changes in sensation, perception, cognition, affect, mood, or behavior.

This study will examine whether or not hypnosis is helpful in reducing breast cancer survivors' AI-related MSP and in improving their adherence to their prescribed AI regimen. This study will also examine whether the hypnosis intervention is cost effective. To answer these questions, this randomized clinical trial will compare hypnosis (three sessions) to a non-hypnosis, attention control, empathic listening condition (three sessions). For each intervention, the first session will be approximately 40 minutes, and sessions 2 and 3 will be approximately 30 minutes each. Both interventions will be delivered face-to-face, by a doctoral-level psychology professional.

All participants will be taking AIs for breast cancer, will be experiencing some musculoskeletal pain since starting AIs (≥3 on a 10 point scale), and will be randomized to one of the two intervention groups. Study participants will be asked to complete measures of pain, AI adherence, and other behavioral and psychosocial measures over the course of 12-month period. The follow-up assessments will evaluate the clinical efficacy and cost-effectiveness of hypnosis versus professional attention.

Overall, this project is a critical step towards reducing the struggles of breast cancer survivors experiencing AI-related MSP, and associated non-adherence. By reducing MSP and improving AI adherence, the hypnosis intervention tested here has the potential to improve quality of life and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosed with Stage 0-III hormone-receptor positive breast cancer
* Taking a third-generation aromatase inhibitor (AI) (e.g., anastrozole (Arimidex), letrozole (Femara), or exemestane (Aromasin)) for at least 3 months left in their AI prescription to complete all study assessments (e.g., at least one year left on AIs)
* Experiencing ongoing pain and/or stiffness in one or more joints, which started or worsened after initiation of AI therapy
* Having a baseline worst pain score over the past week on the Brief Pain Inventory-Short Form (BPI-SF) of ≥ 3 on a 0 to 10 scale
* Over age 18
* Able to speak and read English (to allow for participation in study intervention sessions)
* Consent to the study
* Be willing to be randomized to experimental conditions
* Willing to travel to Mount Sinai for study procedures (e.g., intervention sessions, follow-up appointments).

Exclusion Criteria:

* Inflammatory, metabolic or neuropathic arthropathies at the time of recruitment
* Fibromyalgia
* Past cancer. Patients will be excluded if they have ever been diagnosed with cancer (including DCIS/LCIS) prior to the breast cancer for which the present course of AIs is being prescribed. However, patients will be eligible if they have a history of non-metastatic, non-melanomatous skin cancer
* Metastatic (Stage IV) breast cancer, as their treatment and outcomes typically follow a different course
* Bone fracture/surgery of an extremity during the preceding 6 months
* Non-steroidal joint injection within the last 3 months.
* Current use of corticosteroids, defined as oral, intravenous (IV), or injections of corticosteroids in the past 4 weeks
* Regular use of narcotics.
* Patients will be excluded due to the presence of the following psychiatric conditions: dementia, psychosis, current mania or uncontrolled major depressive disorder, or addictive disorder or current intoxication.
* In the rare instance of the presence of a comorbidity that does not fall into any of the above mentioned exclusion criteria, but that is clinically determined to significantly interfere with the patient's ability to participate in the study (e.g., cognitive impairment)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2016-03; Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Patient-reported musculoskeletal pain (MSP) as measured by the Brief Pain Inventory-Short Form (BPI-SF) | 12 months
  The Brief Pain Inventory-Short Form (BPI-SF) is a self-report questionnaire assessing pain.

SECONDARY OUTCOMES:
eCap measure | 12 months
  Adherence to aromatase inhibitors as measured by the eCap system. The eCap system is a medication event monitoring system that tracks medication usage without active patient input. eCaps record the date and time whenever the cap is opened to remove a pill.
The Australian/Canadian Osteoarthritis Hand Index (AUSCAN) | 12 months
  AUSCAN is a self-report measure of musculoskeletal pain.
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 12 months
  WOMAC is a self-report measure of musculoskeletal pain.
The Breast Cancer Prevention Trial-Musculoskeletal Symptom (BCPT-MS) | 12 months
  BCPT-MS is a self-report measure of musculoskeletal pain.
The Medication Adherence Report Scale (MARS) | 12 months
  MARS is a self-reported measure of AI adherence.
The Healthcare Consumption, Illness and Work Questionnaire (Adapted TiC-P) | 12 months
  Adapted TiC-P is a self-report measure to calculate costs associated with AI-related musculoskeletal pain.

CONTACTS AND LOCATIONS:
Overall Officials: Guy H Montgomery, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

DOCUMENTS (1):
  • Informed Consent Form (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT02657993/ICF_000.pdf